CLINICAL TRIAL: NCT04520256
Title: Rapid Evaluation of Innovative Intervention Components to Maximize the Health Benefits of Behavioral Obesity Treatment Delivered Online: An Application of Multiphase Optimization Strategy
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: R01DK117857 (NIH); R01DK117857 (NIH)
Record Dates: First submitted 2020-08-12; First posted 2020-08-20 (Actual); Results first posted 2025-01-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2024-03

CONDITIONS: Overweight and Obesity
Keywords: Diet; Physical activity; Online
MeSH Terms: conditions — Overweight; Obesity; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (32):
- Core Program Only (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program
- Social Support (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Platform for Social Support & Friendly Competition
- Dysregulated Eating (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Skills Training for Dysregulated Eating
- Social Support, Dysregulated Eating (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Skills Training for Dysregulated Eating; Behavioral: Platform for Social Support & Friendly Competition
- Exercise (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Intervention for Structured Physical Activity
- Social Support, Exercise (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Platform for Social Support & Friendly Competition
- Dysregulated Eating, Exercise (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Skills Training for Dysregulated Eating
- Social Support, Dysregulated Eating, Exercise (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Skills Training for Dysregulated Eating; Behavioral: Platform for Social Support & Friendly Competition
- Feedback (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Interactive Video Feedback
- Social Support, Feedback (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Interactive Video Feedback; Behavioral: Platform for Social Support & Friendly Competition
- Dysregulated Eating, Feedback (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Interactive Video Feedback; Behavioral: Skills Training for Dysregulated Eating
- Social Support, Dysregulated Eating, Feedback (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Interactive Video Feedback; Behavioral: Skills Training for Dysregulated Eating; Behavioral: Platform for Social Support & Friendly Competition
- Exercise, Feedback (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Interactive Video Feedback
- Social Support, Exercise, Feedback (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Interactive Video Feedback; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Platform for Social Support & Friendly Competition
- Dysregulated Eating, Exercise, Feedback (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Interactive Video Feedback; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Skills Training for Dysregulated Eating
- Social Support, Dysregulated Eating, Exercise, Feedback (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Tailored Interactive Video Feedback; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Skills Training for Dysregulated Eating; Behavioral: Platform for Social Support & Friendly Competition
- VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training
- Social Support, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Platform for Social Support & Friendly Competition
- Dysregulated Eating, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Skills Training for Dysregulated Eating
- Social Support, Dysregulated Eating, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Skills Training for Dysregulated Eating; Behavioral: Platform for Social Support & Friendly Competition
- Exercise, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Intervention for Structured Physical Activity
- Social Support, Exercise, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Platform for Social Support & Friendly Competition
- Dysregulated Eating, Exercise, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Skills Training for Dysregulated Eating
- Social Support, Dysregulated Eating, Exercise, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Skills Training for Dysregulated Eating; Behavioral: Platform for Social Support & Friendly Competition
- Feedback, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Interactive Video Feedback
- Social Support, Feedback, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Interactive Video Feedback; Behavioral: Platform for Social Support & Friendly Competition
- Dysregulated Eating, Feedback, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Interactive Video Feedback; Behavioral: Skills Training for Dysregulated Eating
- Social Support, Dysregulated Eating, Feedback, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Interactive Video Feedback; Behavioral: Skills Training for Dysregulated Eating; Behavioral: Platform for Social Support & Friendly Competition
- Exercise, Feedback, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Interactive Video Feedback; Behavioral: Tailored Intervention for Structured Physical Activity
- Social Support, Exercise, Feedback, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Interactive Video Feedback; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Platform for Social Support & Friendly Competition
- Dysregulated Eating, Exercise, Feedback, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Interactive Video Feedback; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Skills Training for Dysregulated Eating
- Social Support, Dysregulated Eating, Exercise, Feedback, VR (Experimental)
  Interventions: Behavioral: Online Behavioral Weight Loss Program; Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training; Behavioral: Tailored Interactive Video Feedback; Behavioral: Tailored Intervention for Structured Physical Activity; Behavioral: Skills Training for Dysregulated Eating; Behavioral: Platform for Social Support & Friendly Competition

INTERVENTIONS:
Behavioral: Online Behavioral Weight Loss Program — A self-guided, online program that helps participants reduce energy intake and gradually increase physical activity.
Behavioral: Virtual Reality for Behavioral Weight Loss Skills Training — This program allows participants to practice behavioral weight loss skills using an online virtual reality system accessed via a Web browser.
  Arms: Dysregulated Eating, Exercise, Feedback, VR; Dysregulated Eating, Exercise, VR; Dysregulated Eating, Feedback, VR; Dysregulated Eating, VR; Exercise, Feedback, VR; Exercise, VR; Feedback, VR; Social Support, Dysregulated Eating, Exercise, Feedback, VR; Social Support, Dysregulated Eating, Exercise, VR; Social Support, Dysregulated Eating, Feedback, VR; Social Support, Dysregulated Eating, VR; Social Support, Exercise, Feedback, VR; Social Support, Exercise, VR; Social Support, Feedback, VR; Social Support, VR; VR
Behavioral: Tailored Interactive Video Feedback — Video-recorded messages are used to provide periodic feedback on progress with weight loss, dietary change, and physical activity. Additional videos provide dietary skills training.
  Arms: Dysregulated Eating, Exercise, Feedback; Dysregulated Eating, Exercise, Feedback, VR; Dysregulated Eating, Feedback; Dysregulated Eating, Feedback, VR; Exercise, Feedback; Exercise, Feedback, VR; Feedback; Feedback, VR; Social Support, Dysregulated Eating, Exercise, Feedback; Social Support, Dysregulated Eating, Exercise, Feedback, VR; Social Support, Dysregulated Eating, Feedback; Social Support, Dysregulated Eating, Feedback, VR; Social Support, Exercise, Feedback; Social Support, Exercise, Feedback, VR; Social Support, Feedback; Social Support, Feedback, VR
Behavioral: Tailored Intervention for Structured Physical Activity — Periodic self-assessment is used to guide selection of a physical activity goal. Home-based instructional videos are provided to help meet the selected goal.
  Arms: Dysregulated Eating, Exercise; Dysregulated Eating, Exercise, Feedback; Dysregulated Eating, Exercise, Feedback, VR; Dysregulated Eating, Exercise, VR; Exercise; Exercise, Feedback, VR; Exercise, VR; Social Support, Dysregulated Eating, Exercise; Social Support, Dysregulated Eating, Exercise, Feedback; Social Support, Dysregulated Eating, Exercise, Feedback, VR; Social Support, Dysregulated Eating, Exercise, VR; Social Support, Exercise; Social Support, Exercise, Feedback; Social Support, Exercise, Feedback, VR; Social Support, Exercise, VR
Behavioral: Skills Training for Dysregulated Eating — Periodic self-assessment is used to guide selection of skills training modules designed to counter common causes of dysregulated eating (e.g., boredom, stress).
  Arms: Dysregulated Eating; Dysregulated Eating, Exercise; Dysregulated Eating, Exercise, Feedback; Dysregulated Eating, Exercise, Feedback, VR; Dysregulated Eating, Exercise, VR; Dysregulated Eating, Feedback; Dysregulated Eating, Feedback, VR; Dysregulated Eating, VR; Social Support, Dysregulated Eating; Social Support, Dysregulated Eating, Exercise; Social Support, Dysregulated Eating, Exercise, Feedback; Social Support, Dysregulated Eating, Exercise, Feedback, VR; Social Support, Dysregulated Eating, Exercise, VR; Social Support, Dysregulated Eating, Feedback; Social Support, Dysregulated Eating, Feedback, VR; Social Support, Dysregulated Eating, VR
Behavioral: Platform for Social Support & Friendly Competition — An online platform is provided for participants to connect with each other, support each other, and compete on achievement of behavioral and weight loss milestones.
  Arms: Social Support; Social Support, Dysregulated Eating; Social Support, Dysregulated Eating, Exercise; Social Support, Dysregulated Eating, Exercise, Feedback; Social Support, Dysregulated Eating, Exercise, Feedback, VR; Social Support, Dysregulated Eating, Exercise, VR; Social Support, Dysregulated Eating, Feedback; Social Support, Dysregulated Eating, Feedback, VR; Social Support, Dysregulated Eating, VR; Social Support, Exercise; Social Support, Exercise, Feedback; Social Support, Exercise, Feedback, VR; Social Support, Exercise, VR; Social Support, Feedback; Social Support, Feedback, VR; Social Support, VR

SUMMARY:
When delivered online, behavioral obesity treatments have the potential to reach large numbers of individuals with overweight/obesity and produce significant improvements in health and wellbeing. In order to maximize the public health benefit of disseminating these treatments online, this study will use the Multiphase Optimization Strategy (MOST) framework to most quickly and efficiently determine which, if any, of 5 innovative intervention components, alone or in combination, increases the proportion of patients achieving a ≥5% weight loss, and mean weight loss, after a 12-month online behavioral obesity treatment.

DETAILED DESCRIPTION:
Decades of research have demonstrated that behavioral obesity treatments can produce clinically significant weight losses that improve health and disease risk/severity. However, these treatments have not been disseminated widely due to high costs and lack of qualified providers. The investigators therefore aim to develop and test a fully automated online obesity treatment that would produce clinically significant weight losses (i.e., ≥ 5 % of initial body weight) when delivered online. In order to maximize the public health impact of online obesity treatment, and advance the science of online behavioral intervention in general, it is imperative to evaluate innovative behavioral intervention components with the potential to optimize weight loss outcomes. Because digital health technology evolves rapidly, this research will use the Multiphase Optimization Strategy (MOST) framework to most quickly and efficiently determine which, if any, of 5 innovative intervention components, alone or in combination, increases the proportion of patients achieving a ≥5% weight loss, and mean weight loss, of the online Rx Weight loss (RxWL) program at 12- months. The 5 intervention components to be tested are: (a) Web-based virtual reality intervention for training in basic behavioral weight loss skills; tailored interactive intervention targeting (b) structured physical activity and (c) dysregulated eating; (d) a platform for social interaction including opportunities for friendly competition, and (e) interactive video feedback with content tailored to the unique needs of each participant and a focus on dietary skills. A sample of 384 individuals with BMI ≥ 25 will be randomized to receive RxWL and 0-5 of the experimental intervention components in a full factorial experiment. This design will allow the investigators to determine which intervention components maximize weight loss and whether there are favorable combinations of components. In addition, by evaluating the effects of each component on proximal outcomes (i.e., mediators) it will be possible learn not only which components are (or are not) effective but also why or how they exert their effects. This project advances the science of behavioral obesity treatment, and will directly impact the care of patients receiving RxWL.

ELIGIBILITY:
* English language fluent and literate at the 6th grade level
* Body mass index (BMI) between 25 and 50 kg/m-squared
* Able to walk 2 city blocks without stopping
* Not currently participating in another weight loss program
* Not currently taking weight loss medication
* Has not lost ≥5% of body weight in the 6 months prior to enrolling
* Has not been pregnant within the 6 months prior to enrolling
* Does not plan to become pregnant within 12 months of enrolling
* Denies having a heart condition, chest pain during periods of activity or rest, or loss of consciousness in the 12 months prior to enrolling
* Denies any medical condition that would affect the safety of participating in unsupervised physical activity
* Denies any condition that would result in inability to follow the study protocol, including terminal illness, substance abuse, eating disorder (not including Binge Eating Disorder) and untreated major psychiatric illness

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 384 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2023-05-18 (Actual); Study Completion 2023-05-18 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Miriam Hospital Weight Control and Diabetes Resarch Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thomas JG, Goldstein CM, Bond DS, Lillis J, Hekler E, Goldstein SP, Butryn ML, Cao Z, Wing RR. Evaluation of Five Novel Intervention Components in Online Obesity Treatment: Outcomes of a Randomized Factorial Experiment. Obesity (Silver Spring). 2025 Nov;33(11):2128-2138. doi: 10.1002/oby.70039. Epub 2025 Sep 18. PMID 40968617

RESULTS

PARTICIPANT FLOW:
Groups:
- Virtual Reality: Online Behavioral Weight Loss Program: A self-guided, online program that helps participants reduce energy intake and gradually increase physical activity.
  Virtual Reality for Behavioral Weight Loss Skills Training: This program allows participants to practice behavioral weight loss skills using an online virtual reality system accessed via a Web browser.
Period: Overall Study
Arm/Group | Core Program Only | Social Support | Dysregulated Eating | Social Support, Dysregulated Eating | Exercise | Social Support, Exercise | Dysregulated Eating, Exercise | Social Support, Dysregulated Eating, Exercise | Feedback | Social Support, Feedback | Dysregulated Eating, Feedback | Social Support, Dysregulated Eating, Feedback | Exercise, Feedback | Social Support, Exercise, Feedback | Dysregulated Eating, Exercise, Feedback | Social Support, Dysregulated Eating, Exercise, Feedback | Virtual Reality | Social Support, VR | Dysregulated Eating, VR | Social Support, Dysregulated Eating, VR | Exercise, VR | Social Support, Exercise, VR | Dysregulated Eating, Exercise, VR | Social Support, Dysregulated Eating, Exercise, VR | Feedback, VR | Social Support, Feedback, VR | Dysregulated Eating, Feedback, VR | Social Support, Dysregulated Eating, Feedback, VR | Exercise, Feedback, VR | Social Support, Exercise, Feedback, VR | Dysregulated Eating, Exercise, Feedback, VR | Social Support, Dysregulated Eating, Exercise, Feedback, VR
Started | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12
Completed | 6 | 8 | 10 | 9 | 6 | 6 | 8 | 6 | 11 | 9 | 9 | 10 | 7 | 9 | 9 | 6 | 6 | 8 | 9 | 9 | 5 | 9 | 9 | 4 | 7 | 8 | 9 | 8 | 9 | 8 | 8 | 8
Not Completed | 6 | 4 | 2 | 3 | 6 | 6 | 4 | 6 | 1 | 3 | 3 | 2 | 5 | 3 | 3 | 6 | 6 | 4 | 3 | 3 | 7 | 3 | 3 | 8 | 5 | 4 | 3 | 4 | 3 | 4 | 4 | 4
Not completed — Lost to Follow-up | 6 | 4 | 2 | 3 | 6 | 6 | 4 | 6 | 1 | 3 | 3 | 2 | 5 | 3 | 3 | 6 | 6 | 4 | 3 | 3 | 7 | 3 | 3 | 8 | 5 | 4 | 3 | 4 | 3 | 4 | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Core Program Only | Social Support | Dysregulated Eating | Social Support, Dysregulated Eating | Exercise | Social Support, Exercise | Dysregulated Eating, Exercise | Social Support, Dysregulated Eating, Exercise | Feedback | Social Support, Feedback | Dysregulated Eating, Feedback | Social Support, Dysregulated Eating, Feedback | Exercise, Feedback | Social Support, Exercise, Feedback | Dysregulated Eating, Exercise, Feedback | Social Support, Dysregulated Eating, Exercise, Feedback | Virtual Reality | Social Support, VR | Dysregulated Eating, VR | Social Support, Dysregulated Eating, VR | Exercise, VR | Social Support, Exercise, VR | Dysregulated Eating, Exercise, VR | Social Support, Dysregulated Eating, Exercise, VR | Feedback, VR | Social Support, Feedback, VR | Dysregulated Eating, Feedback, VR | Social Support, Dysregulated Eating, Feedback, VR | Exercise, Feedback, VR | Social Support, Exercise, Feedback, VR | Dysregulated Eating, Exercise, Feedback, VR | Social Support, Dysregulated Eating, Exercise, Feedback, VR | Total
Number analyzed (Participants) | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 384
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.5 (10.8) | 54.3 (11.8) | 53.6 (11.9) | 53.6 (8.9) | 58.3 (8.5) | 48 (11.3) | 56.2 (11.0) | 57.7 (9.1) | 53.3 (12.7) | 46.7 (13.0) | 56.3 (10.2) | 52.2 (13.5) | 52.9 (12.6) | 58.6 (9.9) | 56 (12.7) | 50.8 (11.6) | 53.3 (12.3) | 54.9 (7.4) | 56.8 (13.2) | 50.0 (13.2) | 55.4 (10.6) | 57.1 (12.4) | 58.2 (11.5) | 55 (9.1) | 51.5 (11.7) | 51.9 (9.3) | 52 (13.3) | 51.2 (14.0) | 49.6 (16.7) | 49.3 (10.1) | 53.9 (12.3) | 44.5 (13.4) | 53.4 (12.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 2 | 0 | 2 | 2 | 1 | 1 | 2 | 2 | 2 | 2 | 1 | 1 | 2 | 4 | 0 | 1 | 1 | 2 | 1 | 2 | 2 | 1 | 2 | 2 | 3 | 1 | 0 | 3 | 1 | 2 | 1 | 1 | 50
  Female | 8 | 12 | 10 | 8 | 10 | 10 | 10 | 10 | 10 | 10 | 11 | 11 | 10 | 8 | 12 | 10 | 11 | 10 | 11 | 8 | 10 | 11 | 10 | 10 | 7 | 11 | 12 | 9 | 11 | 9 | 10 | 10 | 320
  Other | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 3
  Unknown or Not Reported | 2 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 2 | 0 | 1 | 0 | 2 | 1 | 1 | 0 | 0 | 1 | 2 | 2 | 1 | 20
  Not Hispanic or Latino | 10 | 11 | 10 | 10 | 11 | 11 | 12 | 11 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 10 | 12 | 11 | 11 | 8 | 12 | 11 | 12 | 7 | 11 | 11 | 12 | 12 | 11 | 10 | 9 | 10 | 350
  Unknown or Not Reported | 2 | 1 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 1 | 0 | 0 | 1 | 1 | 00 | 1 | 2 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 2 | 2 | 0 | 0 | 1 | 1 | 1 | 2 | 4 | 0 | 0 | 2 | 1 | 2 | 3 | 38
  White | 7 | 11 | 9 | 11 | 10 | 8 | 6 | 11 | 11 | 8 | 10 | 12 | 11 | 11 | 11 | 8 | 11 | 9 | 9 | 10 | 12 | 10 | 11 | 7 | 8 | 7 | 12 | 11 | 9 | 10 | 9 | 8 | 308
  More than one race | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 9
  Unknown or Not Reported | 2 | 0 | 1 | 1 | 1 | 3 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 22
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 12 | 384

OUTCOME MEASURES:

1. Primary Outcome: Weight Change (Percent of Initial Body Weight) From Baseline to Month 12, Main Effect of Time
Description: Weight was measured at the research center by the research team, or measured by the participant at home and sent to the research team with with documentation of the value reported (e.g., a photograph from a home scale showing the weight).
  A change between two time points is reported. The value of this outcome was calculated using: [(baseline weight - month 12 weight) ÷ baseline weight] × 100. Estimated mean change was obtained from a linear mixed models analysis of variance. Data from all randomized participants were included in the model (ITT analysis).
Time Frame: From Baseline to Month 12
Measure: Mean (Standard Error); unit: percent of initial body weight
Groups:
- All Participants: All participants regardless of random assignment to intervention components.
Arm/Group | All Participants
Number analyzed (Participants) | 384
percent of initial body weight | -5.8 (0.87)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p < .001, Mixed Models Analysis

2. Primary Outcome: Weight Change (Percent of Initial Body Weight) From Baseline to Month 12, Time by Intervention Component Interaction
Description: Weight was measured at the research center by the research team, or measured by the participant at home and sent to the research team with with documentation of the value reported (e.g., a photograph from a home scale showing the weight).
  A change between two time points is reported. The value of this outcome was calculated using: [(baseline weight - month 12 weight) ÷ baseline weight] × 100. Estimated mean change was obtained from a linear mixed models analysis of variance. Data from all randomized participants were included in the model (ITT analysis).
  This outcome measure is reported as an additional effect beyond that of Outcome Measure 1 (each intervention component has it's own weight loss effect that is above and beyond the weight change calculated in the Outcome Measure 1 analyses).
Time Frame: From Baseline to Month 12
Population: All randomized participants.
Measure: Mean (Standard Error); unit: percent of initial body weight
Groups:
- Social Support: An online platform is provided for participants to connect with each other, support each other, and compete on achievement of behavioral and weight loss milestones.
- Dysregulated Eating: Periodic self-assessment is used to guide selection of skills training modules designed to counter common causes of dysregulated eating (e.g., boredom, stress).
- Exercise: Periodic self-assessment is used to guide selection of a physical activity goal. Home-based instructional videos are provided to help meet the selected goal.
- Feedback: Video-recorded messages are used to provide periodic feedback on progress with weight loss, dietary change, and physical activity. Additional videos provide dietary skills training.
- Virtual Reality: This program allows participants to practice behavioral weight loss skills using an online virtual reality system accessed via a Web browser.
Arm/Group | Social Support | Dysregulated Eating | Exercise | Feedback | Virtual Reality
Number analyzed (Participants) | 384 | 384 | 384 | 384 | 384
percent of initial body weight | -0.27 (0.70) | 0.09 (0.70) | -0.03 (0.70) | 0.44 (0.70) | 0.92 (0.70)
Statistical Analysis 1: Comparison: Social Support; Test type: Superiority; p = 0.693, Mixed Models Analysis; Estimated Change = -0.27, 95% CI 2-sided [-.54 to 0.01]
Statistical Analysis 2: Comparison: Dysregulated Eating; Test type: Superiority; p = 0.900, Mixed Models Analysis; Estimated Change = 0.09, 95% CI 2-sided [0.01 to 0.18]
Statistical Analysis 3: Comparison: Exercise; Test type: Superiority; p = 0.960, Mixed Models Analysis; Estimated Change = -0.03, 95% CI 2-sided [-0.06 to 0.01]
Statistical Analysis 4: Comparison: Feedback; Test type: Superiority; p = 0.113, Mixed Models Analysis; Estimated Change = 0.44, 95% CI 2-sided [0.01 to 0.88]
Statistical Analysis 5: Comparison: Virtual Reality; Test type: Superiority; p = 0.187, Mixed Models Analysis; Estimated Change = 0.92, 95% CI 2-sided [0.01 to 1.84]

3. Primary Outcome: Proportion of Participants With Weight Loss ≥ 5% at Month 12, Main Effect of Time
Description: Weight was measured at the research center by the research team, or measured by the participant at home and sent to the research team with with documentation of the value reported (e.g., a photograph from a home scale showing the weight).
  Weight loss was calculated using: [(baseline weight - month 12 weight) ÷ baseline weight] × 100.
  The estimated proportion of participants achieving a weight loss of ≥ 5% of their Baseline body weight was obtained from a generalized linear mixed models analysis of variance to account for missing data. All randomized participants were utilized in the model (ITT analysis).
Time Frame: Month 12
Measure: Mean (Standard Error); unit: proportion of participants
Arm/Group | All Participants
Number analyzed (Participants) | 384
proportion of participants | 0.08 (0.15)
Statistical Analysis 1: Comparison: All Participants; Test type: Superiority; p = 0.999, Mixed Models Analysis

4. Primary Outcome: Proportion of Participants With Weight Loss ≥ 5% at Month 12, Time by Intervention Component Interaction
Description: Weight was measured at the research center by the research team, or measured by the participant at home and sent to the research team with with documentation of the value reported (e.g., a photograph from a home scale showing the weight).
  Weight loss was calculated using: [(baseline weight - month 12 weight) ÷ baseline weight] × 100.
  Estimated proportions of participants with weight loss of ≥ 5% of initial body weight at Month 12 were obtained from a generalized linear mixed models analysis of variance to account for missing data. All randomized participants were utilized in the model (ITT analysis).
Time Frame: Month 12
Population: All randomized participants.
Measure: Mean (Standard Error); unit: proportion of participants
Arm/Group | Social Support | Dysregulated Eating | Exercise | Feedback | Virtual Reality
Number analyzed (Participants) | 384 | 384 | 384 | 384 | 384
proportion of participants | .12 (.23) | .15 (.27) | .11 (.21) | .11 (.20) | .10 (.19)
Statistical Analysis 1: Comparison: Social Support; Test type: Superiority; p = .999, Mixed Models Analysis; Estimated Proportion = .12, 95% CI 2-sided [0 to .56]
Statistical Analysis 2: Comparison: Dysregulated Eating; Test type: Superiority; p = .999, Mixed Models Analysis; Estimated Proportion = .15, 95% CI 2-sided [0 to .68]
Statistical Analysis 3: Comparison: Exercise; Test type: Superiority; p = .999, Mixed Models Analysis; Estimated Proportion = .11, 95% CI 2-sided [0 to .52]
Statistical Analysis 4: Comparison: Feedback; Test type: Superiority; p = .999, Mixed Models Analysis; Estimated Proportion = .11, 95% CI 2-sided [0 to .50]
Statistical Analysis 5: Comparison: Virtual Reality; Test type: Superiority; p = .999, Mixed Models Analysis; Estimated Proportion = .10, 95% CI 2-sided [0 to .47]

ADVERSE EVENTS:
Time Frame: 12 months from Baseline
Arm/Group | Core Program Only | Social Support | Dysregulated Eating | Social Support, Dysregulated Eating | Exercise | Social Support, Exercise | Dysregulated Eating, Exercise | Social Support, Dysregulated Eating, Exercise | Feedback | Social Support, Feedback | Dysregulated Eating, Feedback | Social Support, Dysregulated Eating, Feedback | Exercise, Feedback | Social Support, Exercise, Feedback | Dysregulated Eating, Exercise, Feedback | Social Support, Dysregulated Eating, Exercise, Feedback | Virtual Reality | Social Support, VR | Dysregulated Eating, VR | Social Support, Dysregulated Eating, VR | Exercise, VR | Social Support, Exercise, VR | Dysregulated Eating, Exercise, VR | Social Support, Dysregulated Eating, Exercise, VR | Feedback, VR | Social Support, Feedback, VR | Dysregulated Eating, Feedback, VR | Social Support, Dysregulated Eating, Feedback, VR | Exercise, Feedback, VR | Social Support, Exercise, Feedback, VR | Dysregulated Eating, Exercise, Feedback, VR | Social Support, Dysregulated Eating, Exercise, Feedback, VR
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/56/NCT04520256/Prot_SAP_000.pdf